CLINICAL TRIAL: NCT03475901
Title: A Feasibility Study for the Use of Virtual Reality to Reduce Procedural Anxiety for Children Undergoing Laceration Repair in the Pediatric Emergency Room
Brief Title: Virtual Reality for Anxiolysis During Laceration Repair in the Pediatric Emergency Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: KindVR (Unknown)
Responsible Party: Principal Investigator, Daniel Marc Fein, Assistant Professor of Pediatrics, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-8466
Record Dates: First submitted 2018-03-10; First posted 2018-03-23 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Procedural Anxiety; Laceration of Skin
Keywords: procedural anxiety; virtual reality; anxiolysis; laceration repair; pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtualy Reality App (Experimental): Virtual reality app produced by KindVR played via a stereoscopic head mounted display (Samsung GearVR) and headphones that the patient will wear over their eyes and ears.
  Interventions: Other: Virtual Reality App

INTERVENTIONS:
Other: Virtual Reality App — Virtual reality app produced by KindVR played via a stereoscopic head mounted display (Samsung GearVR) and headphones that the patient will wear over their eyes and ears.

SUMMARY:
The investigators propose a pilot study to examine the feasibility of utilizing immersive virtual reality to reduce procedural anxiety in children undergoing non-facial laceration repair in the Pediatric Emergency Department.

The investigators hypothesize that virtual reality will be well-received by patients and their caregivers, and that the anxiety provoked by laceration repair will be mitigated by the immersive virtual reality experience.

ELIGIBILITY:
Inclusion Criteria:

* children 5-13 years of age
* present to ED during the study period with non-facial lacerations
* patient to undergo wound closure with sutures

Exclusion Criteria:

* Patients with lacerations on the head/face
* Patients with lacerations sustained in conjunction with loss of consciousness, altered mental status, life-threatening injuries/illness or multi-trauma
* Patients who sustained a laceration in conjunction with an open fracture
* Patients with open skin, lice, scabies, or other infectious skin conditions on the head/face
* Patients with a history of or current symptoms of vertigo
* Patients who are blind
* Patients with significant developmental or cognitive delays who may not be able to engage with or tolerate the virtual reality environment, as determined by their parent/caregiver
* Patients on whom the VR headset does not fit appropriately
* Non-English speaking patients will be excluded from this study (we do not have funds available to translate the study documents into other languages)

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
The percentage of children whose anxiety score did NOT increase by ≥ 20mm on a visual analog anxiety scale | from the time of enrollment to the placement of the first stitch, which is typically ranges from 15 to 90 minutes
  Anxiety score will be measured on a Visual Analog Scale. This scale consists of a 100mm line on which parents mark their estimate of their child's anxiety level, with anxiety level increasing from left (0mm) to right (100mm).

SECONDARY OUTCOMES:
Change in anxiety score | from the time of enrollment to wound irrigation, which typically ranges from 5 to 80 minutes
  Anxiety score will be measured on a Visual Analog Scale. This scale consists of a 100mm line on which parents mark their estimate of their child's anxiety level, with anxiety level increasing from left (0mm) to right (100mm).
Change in anxiety score | from enrollment to local/regional anesthesia, which typically ranges from 15 to 100 minutes
  Anxiety score will be measured on a Visual Analog Scale. This scale consists of a 100mm line on which parents mark their estimate of their child's anxiety level, with anxiety level increasing from left (0mm) to right (100mm).
Change in anxiety score | from enrollment to procedure completion, which typically ranges from 20 to 180 minutes
  Anxiety score will be measured on a Visual Analog Scale. This scale consists of a 100mm line on which parents mark their estimate of their child's anxiety level, with anxiety level increasing from left (0mm) to right (100mm).
Patient satisfaction with the use of VR during the procedure as assessed by a patient questionnaire | Patients will fill out the questionnaire at the time their sutured laceration repair is completed, which is typically between 20 and 180 minutes after enrollment
  To assess the receptiveness of patients to this technology as well as the efficacy of the VR experience, participants will be asked to complete a brief questionnaire at the end of the procedure assessing their experience while using VR during the laceration repair.
  These surveys address the patient's comfort and satisfaction with the technology. We have created separate patient surveys for children ages 5-7 and children ages 8-13 - these surveys have the same questions, but the answer choices are simplified from Likert Rating Scales (scale of 1 - 5) for the older children to a simple "Yes, No, I don't know" choice for the younger children. There is also a free text response question for which patients can provide additional comments or suggestions regarding their use of VR during laceration repair.
Parent/guardian satisfaction with the use of VR during the procedure as assessed by a parent/guardian questionnaire | Parent/guardian will fill out the questionnaire at the time their child's sutured laceration repair is completed, which is typically between 20 and 180 minutes after enrollment
  To assess the receptiveness of patients to this technology as well as the efficacy of the VR experience, parents/guardians will be asked to complete a brief survey at the end of the procedure assessing their comfort and satisfaction with their child's use of VR during the laceration repair. The survey contains both rating questions with Likert Rating Scales (scale of 1 - 5), yes/no questions, and questions with free text responses.
Provider satisfaction with the use of VR during the procedure as measured by a provider questionnaire | Providers will fill out the questionnaire at the time their patient's sutured laceration repair is completed, which is typically between 20 and 180 minutes after enrollment
  The ED provider who performed the laceration repair will complete a survey at the end of the procedure assessing their satisfaction with using VR during laceration repair. The survey contains yes/no questions, multiple choice questions, and questions with free text responses.
Need for adjunctive anxiolysis methods, sedation, or restraints during the procedure as reported on a provider questionnaire | from enrollment to procedure completion, which typically ranges from 20 to 180 minutes
  The ED provider who performed the laceration repair will complete a questionnaire at the end of the procedure which will detail which, if any, adjunctive measures were needed during the procedure.
Headache due to VR use as reported on a qualitative simulator sickness questionnaire | from enrollment to procedure completion, which typically ranges from 20 to 180 minutes
  The patient (with the help of their parent/guardian for younger children) will complete a questionnaire assessing for symptoms of simulator sickness, including nausea, headache, dizziness, and eye pain. The questionnaire uses Likert Scales (ranging from 1 to 5, with 5 indicating a higher level of symptom) to assess nausea, headache, dizziness, and eye pain associated with VR use.
Eye pain due to VR use as reported on a qualitative simulator sickness questionnaire | from enrollment to procedure completion, which typically ranges from 20 to 180 minutes
  The patient (with the help of their parent/guardian for younger children) will complete a questionnaire assessing for symptoms of simulator sickness, including nausea, headache, dizziness, and eye pain. The questionnaire uses Likert Scales (ranging from 1 to 5, with 5 indicating a higher level of symptom) to assess nausea, headache, dizziness, and eye pain associated with VR use.
Nausea due to VR use as reported on a qualitative simulator sickness questionnaire | from enrollment to procedure completion, which typically ranges from 20 to 180 minutes
  The patient (with the help of their parent/guardian for younger children) will complete a questionnaire assessing for symptoms of simulator sickness, including nausea, headache, dizziness, and eye pain. The questionnaire uses Likert Scales (ranging from 1 to 5, with 5 indicating a higher level of symptom) to assess nausea, headache, dizziness, and eye pain associated with VR use.
Dizziness due to VR use as reported on a qualitative simulator sickness questionnaire | from enrollment to procedure completion, which typically ranges from 20 to 180 minutes
  The patient (with the help of their parent/guardian for younger children) will complete a questionnaire assessing for symptoms of simulator sickness, including nausea, headache, dizziness, and eye pain. The questionnaire uses Likert Scales (ranging from 1 to 5, with 5 indicating a higher level of symptom) to assess nausea, headache, dizziness, and eye pain associated with VR use.
Barriers to the use of VR identified during this study as reported on a provider questionnaire | from enrollment to procedure completion, which typically ranges from 20 to 180 minutes
  The ED provider who performed the laceration repair will complete a questionnaire at the end of the procedure which will detail which, if any, barriers to the use of VR that they encountered during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Fein, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Children's Hospital at Montefiore, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nemetski SM, Berman DI, Khine H, Fein DM. Virtual Reality as Anxiolysis During Laceration Repair in the Pediatric Emergency Department. J Emerg Med. 2022 Jul;63(1):72-82. doi: 10.1016/j.jemermed.2022.01.025. Epub 2022 Aug 5. PMID 35934650